CLINICAL TRIAL: NCT00531882
Title: A Pilot Study Evaluating the Effect of Pioglitazone, Simvastatin, and Ibuprofen on Neutrophil Migration in Vivo in Healthy Subjects
Brief Title: Pilot Mouthwash Study of Pioglitazone and Simvastatin in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Michael W. Konstan, Chairman Department of Pediatrics, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pilot Healthy Volunteers
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Results first posted 2017-07-28 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Cystic Fibrosis
Keywords: healthy volunteers; neutrophil migration; anti inflammatory non-steroidal agent; simvastatin; pioglitazone
MeSH Terms: conditions — Cystic Fibrosis | interventions — Pioglitazone; Simvastatin; Ibuprofen

STUDY DESIGN:
Masking Description: No person associated with the study was masked
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1-pioglitazone (Experimental): Pioglitazone
  Interventions: Drug: Pioglitazone
- 2-simvasatin (Experimental): Simvastatin
  Interventions: Drug: Simvastatin
- 3-Ibuprofen 1000-1600 mg/day (Active Comparator): Ibuprofen 1000-16-- mg/day, maximum 3200 mg/day
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Pioglitazone — 30 mg once a day
  Other Names: ACTOS
  Arms: 1-pioglitazone
Drug: Simvastatin — 40 mg once a day
  Other Names: Zocor
  Arms: 2-simvasatin
Drug: Ibuprofen — Ibuprofen 15-23 mg/kg twice daily, maximum 3200 mg/day
  Other Names: Motrin
  Arms: 3-Ibuprofen 1000-1600 mg/day

SUMMARY:
Inflammation clearly contributes to the progression of the cystic fibrosis (CF) lung disease, and administration of the anti-inflammatory agent high-dose ibuprofen retards the rate of decline of pulmonary function. However, utilization of this valuable drug has been suboptimal because of its rare, but dramatic, adverse effects. Therefore, alternative anti-inflammatory agents are urgently needed. One strategy for identifying new anti-inflammatory agents is to determine the mechanism by which the only proven anti-inflammatory agent for the CF lung disease, high-dose ibuprofen, exerts its effect. If this were known, then other drugs that act by a similar mechanism become candidates for treating the CF inflammatory disease. The investigators have shown, in our preliminary studies, that high dose ibuprofen limits the delivery of neutrophils to an inflamed mucosal surface, the gingival crevices. The investigators plan to test pioglitazone and simvastatin, (ibuprofen (positive control)) to determine their anti inflammatory affects on neutrophil migration to the oral mucosa.

The hypothesis to be tested is that pioglitazone, and/or simvastatin will reduce neutrophils in the oral mucosa after 10 days of therapy in mouthwashes of healthy volunteers. Ibuprofen will be used as a positive control.

This study will provide pilot data from healthy volunteers to support an FDA Grant to be submitted at a future date.

DETAILED DESCRIPTION:
The entire study period for each subject will be 15 days, and consist of 3 periods defined as: Baseline (Day 1,2,3), Treatment (Day 3-10), and Recovery (Day 13-15). Healthy volunteers will be screened on Day 1 (and assessed for eligibility); Eligible subjects will be divided into 3 drug treatment groups pioglitazone, simvastatin and ibuprofen the positive control. The two treatment groups will consist of 4 healthy volunteers who meet the inclusion criteria. There will be 2 healthy volunteers in the positive control group. Group 1 will receive pioglitazone 30 mg once daily, Group 2 will receive simvastatin 40 mg daily and Group 3 the positive control will receive ibuprofen (15-23 mg/kg twice daily, maximum 3200 mg/day) during the Treatment period and serve as the positive control group. This dose is 25% of that prescribed to CF patients. As healthy volunteers are recruited, the first will be assigned to Group 1, the second to Group 2, and so on. After the third subject has been assigned to Group 3, this pattern of assignment will be repeated with subjects 4, 5 and 6, The following 4 healthy volunteers will be assigned to group 1 and 2 (7, 8, 9, 10).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 < 50 years of age
* Healthy volunteers must be in general good health as determined by a medical history.
* Ability to understand and sign the informed consent form
* Ability to adhere to the protocol.
* Willing to use an acceptable form of birth control

Exclusion Criteria:

* History of diabetes requiring insulin
* The use of NSAIDS (ibuprofen) or corticosteroids including inhaled steroids. Nasal steroids are acceptable.
* The use of statin lowering medications
* Active gingival disease (Active tooth or gum disease)
* Any chronic inflammatory condition that immuno compromises the volunteer as determined by medical history.
* Pregnant or planning to become pregnant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2007-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Konstan, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (2):
- United States (2):
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from lab personnel and CF Center employees and UH employees and by word of mouth. Due to the vulnerability of this population every effort was made to avoid coercion. No one was enrolled that was directly supervised by the PI. The recruitment log was kept in a secure location in the CF Team Office.
Pre-assignment Details: Inclusion and exclusion criteria were reviewed at screening. Concomitant medications were reviewed prior to randomization. Subjects were excluded if they were on NSAIDS, corticosteroids (including inhaled steroids and statin lowering medications.
Groups:
- 1-Pioglitazone: Pioglitazone
  Pioglitazone: 30 mg once a day pioglitazone (Actos, Takeda) will be administered orally in a dose of 30 mg once daily. This is the highest recommended dose for initial control of type II diabetes.
- 2-Simvastatin: Simvastatin (Zocor): 40 mg once a day will be administered orally in a dose of 49 mg once daily to all subjects. This dose is considered a mid-level adult dose and the maximum pediatric dose recommended for hyperlipidemia.
- 3-Ibuprofen 1000-1600 mg Twice Daily (Max 3200 mg/Day): Ibuprofen will be used as the positive control for this study. Ibuprofen (Motrin, Pharmacia) will be administered twice daily.
Period: Overall Study
Arm/Group | 1-Pioglitazone | 2-Simvastatin | 3-Ibuprofen 1000-1600 mg Twice Daily (Max 3200 mg/Day)
Started | 10 | 10 | 5
Completed | 10 | 10 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This study was conducted to provide data as proof of concept and to provide pilot data to support an FDA grant to be submitted at a later date.
Groups:
- 2-Simvastin: Simvastatin
  Simvastatin: 40 mg once a day
- 3-Ibuprofen 1000-1600 mg Twice Daily: Ibuprofen 1000-1600 mg twice daily (max 3200 mg/day)
- Total: Total of all reporting groups
Arm/Group | 1-Pioglitazone | 2-Simvastin | 3-Ibuprofen 1000-1600 mg Twice Daily | Total
Number analyzed (Participants) | 10 | 10 | 5 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 5 | 25
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.4 (8.8) | 28.8 (9.1) | 24.5 (4.0) | 27.6 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 3 | 14
  Male | 4 | 5 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Neutrophil Delivery to the Oral Mucosa Using a Non-invasive Mouthwash Technique
Description: Oral mucosal polymorphonuclear leukocytes (PMN) are obtained and assessed using a modification of the mouthwash method of (Wright et.al. Blood 1986;67:1023-30). For each subject, PMN counts are assessed on days 1, 2, 3 [Baseline (B)]; days 8, 9, 10 [Treatment (T)]; and days 11, 13, 15 [Recovery (R)]. The PMN counts for each subject are averaged for each study time period (B, T or R) within each study arm (Pioglitazone, Simvastatin and Ibuprofen). The mean baseline (B) PMN counts are compared to the mean treatment (T) PMN counts for each study arm, with the results expressed as the percent change in PMN counts . Paired T-tests between baseline and treatment PMN counts are used to analyze for significance. The recovery period is used to verify that the PMN counts return to baseline following the treatment period. Data from the recovery period is not shown.
Time Frame: 3X Before treatment (Days 1,2,3) 3X During treatment (Days 8,9,10)
Population: Healthy volunteers free of gingival disease were randomized 2:2:1 to oral Pioglitazone, Simvastatin or Ibuprofen respectively for 10 days.
Measure: Number; unit: % change in mean PMN counts: B vs T
Groups:
- 2-Simvastatin: Simvastatin
  Simvastatin: 40 mg once a day
- 3-Ibuprofen 1000-1600 mg Twice Daily (Max 3200 mg/Day): Ibuprofen 15-23 mg/kg twice daily, maximum 3200 mg/day
  Ibuprofen: Ibuprofen 15-23 mg/kg twice daily, maximum 3200 mg/day
Arm/Group | 1-Pioglitazone | 2-Simvastatin | 3-Ibuprofen 1000-1600 mg Twice Daily (Max 3200 mg/Day)
Number analyzed (Participants) | 10 | 10 | 5
% change in mean PMN counts: B vs T | 6.4 | -19.6 | -28.4

ADVERSE EVENTS:
Time Frame: Subjects were questioned and examined by the Investigator or his/her designee for evidence of adverse events. Subjects were monitored for the 15 days they participated in the study.
Arm/Group | 1-Pioglitazone | 2-Simvastin | 3-Ibuprofen 1000-1600 mg Twice Daily (Max 3200 mg/Day)
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 0/10 | 2/10 | 0/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1-Pioglitazone (N=10) | 2-Simvastin (N=10) | 3-Ibuprofen 1000-1600 mg Twice Daily (Max 3200 mg/Day) (N=5)
joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) — joint pain possibly related to simvastatin

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes